CLINICAL TRIAL: NCT04842422
Title: Earliest Stage Treatment of Aktinic Keratosis With Imiquimod 3.75% Cream
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12020
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Earliest Stage Treatment of Aktinic Keratosis (Experimental)
  Interventions: Drug: Imiquimod 3.75% Cream

INTERVENTIONS:
Drug: Imiquimod 3.75% Cream — Imiquimod 3.75% Cream

SUMMARY:
Earliest Stage Treatment of Actinic Keratosis with Imiquimod 3.75% Cream:

The study is to demonstrate that Aktinic Keratosis are present before they are clinically visible, i.e. in a subclinical stage. Since on the basis of the research situation, also subclinical AK can proliferate into the dermis, it is possible that with the application of Imiquimod on chronically light-exposed skin, undetected squamous cell carcinoma can be recognized and treated at the same time.

ELIGIBILITY:
Inclusion

* Male and female supposed-healthy volunteer outpatients, age: > 50 years.
* Diagnosis: patients with chronically UV-exposed photodamaged facial skin.
* Consent by signing the ICF (Informed Consent Form)

Exclusion

* Current participation in another clinical trial
* Patients who are using topical glucocorticoids on the face.
* Known intolerance/hypersensitivity to imiquimod
* Pregnant/breastfeeding women
* Systemic disease, immunodeficiency

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
immunomodulatory-induced inflammatory reaction | two weeks
  Percentage of subjects in whom an immunomodulatory-induced inflammatory reaction occurs on chronically light-exposed uv-damaged facial skin after two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik für Dermatologie und Venerologie, Graz, Austria